CLINICAL TRIAL: NCT06431633
Title: A Phase III Clinical Trial of Adjuvant Treatment With Sacituzumab and Zimberelimab for Stage IB-IIIA-IIIB(N2) Previously Resected (R0) Non-small Cell Lung Cancer Patients That Did Not Achieve Pathological Complete Response After Neoadjuvant treatment_ARIAN
Brief Title: Study of Treatment With Sacituzumab and Zimberelimab for Patients With Lung Cancer Confined to the Chest and Previously Operated on Who Were Not Disease-free.
Acronym: ARIAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 23/03_ARIAN; 2024-512960-75-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases; Carcinoma, Non-Small-Cell Lung; Resectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Diseases; Carcinoma, Non-Small-Cell Lung | interventions — zimberelimab; sacituzumab govitecan; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM 1: Observation-investigator decision (Active Comparator): Patients randomized in this arm will be in observation for 10 months. It is allowed to administer adjuvant treatment according to investigator criteria. Immunotherapy is not allowed in this arm, only chemotherapy treatment is allowed.
  Interventions: Drug: Cisplatin; Drug: Carboplatin
- ARM 2: Immunotherapy. Zimberelimab treatment for 13 cycles (Experimental): Adjuvant treatment with Zimberelimab will start between the 3rd to the 10th week from surgery. 13 cycles will be administered in total. Cycles will be administered in 21-day intervals (Q3W).
  Zimberelimab: day 1 360 mg IV Q3W (13 cycles)
  Interventions: Drug: Zimberelimab
- ARM 3: Sacituzumab Govitecan + Zimberelimab for 8 cycles + Zimberelimab for 5 cycles (Experimental): Sacituzumab Govitecan: day 1 and 8; 10mg/Kg IV Q3W Zimberelimab: day 1 360 mg IV Q3W
  Treatment sequence:
  Adjuvant treatment will start between the 3rd to the 10th week from surgery. 13 cycles will be administered in total. Cycles will be administered in 21-day intervals (Q3W).
  Patients will receive 8 cycles of Sacituzumab Govitecan + Zimberelimab and 5 cycles of Zimberelimab monotherapy.
  Interventions: Drug: Zimberelimab; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Zimberelimab — Zimberelimab is a fully human IgG4 monoclonal antibody targeting human PD-1. PD-1 is a type I transmembrane protein that is part of the immunoglobulin gene superfamily and the CD28 family of cell surface receptors. PD-1 is an inhibitory immune checkpoint protein that is expressed on activated B cells, T cells, and myeloid cells, and it plays a key role in limiting the activity of effector T cells.
  Zimberelimab is formulated at 30 mg/mL in a buffer solution containing histidine/histidine-HCl buffer solution, sucrose, sodium chloride, and polysorbate 80, at pH 5.5. The investigational product is supplied as a vial contains 120 mg of active Zimberelimab at a concentration of 30mg/mL.
  No premedication nor profilaxis is needed before Zimberelimab administration. Zimberelimab doses are administered by IV infusion over 60 minutes, followed by a 30- to 60-minute observation period, on D1 of each 21-day cycle.
  Other Names: anti-PD-1 monoclonal antibody AB122
  Arms: ARM 2: Immunotherapy. Zimberelimab treatment for 13 cycles; ARM 3: Sacituzumab Govitecan + Zimberelimab for 8 cycles + Zimberelimab for 5 cycles
Drug: Sacituzumab govitecan — Sacituzumab govitecan (SG) is an ADC composed of the following 3 components:
  o The humanized monoclonal antibody hRS7 IgG1κ, which binds to Trop-2, a transmembrane calcium signal transducer that is overexpressed in many epithelial cancers.
  o The camptothecin-derived agent SN-38, a topoisomerase I inhibitor. o A hydrolyzable linker, with the company designation as CL2A that links the humanized monoclonal antibody to SN-38.
  Sacituzumab govitecan is approved globally for the treatment of unresectable locally advanced or metastatic triple-negative breast cancer (TNBC) and HR+ breast cancer.
  Other Names: Trodelvy
  Arms: ARM 3: Sacituzumab Govitecan + Zimberelimab for 8 cycles + Zimberelimab for 5 cycles
Drug: Cisplatin — Cisplatin-based adjuvant chemotherapy
  Cisplatin - CAS 15663-27-1, is a platinum coordination complex with potent anti-neoplastic activity. Induces apoptosis in cancer cells, possibly via caspase-3 activation.
  Other Names: Platinol
  Arms: ARM 1: Observation-investigator decision
Drug: Carboplatin — Cisplatin-based adjuvant chemotherapy Structure: The cis-diamino (cyclobutane-1, 1 dicarboxylate) plating. Stability: 24 hours at ambient temperature in 5% glucose, glucosamine or physiologic saline. It is recommended not to dilute with chlorinated solutions for this could affect the carboplatin. Route of administration: Intravenous infusion. Guidelines of Carboplatin administration: According to the standard of each center. Other Name: ATC code: L01XA02
  Other Names: Paraplatin
  Arms: ARM 1: Observation-investigator decision

SUMMARY:
Open-label, phase III, randomized, stratified (PDL1- vs PDL1+), 3 arms, multicenter clinical trial.

129 resected patients (43 per arm) with stage from IB to IIIA and IIIB (N2) non-small cell lung cancer that do not achieve pathologic complete response (pCR) after neoadjuvant treatment.

This clinical trial has 3 arms of treatment. ARM 1: Observation 10 months, ARM 2: treatment with immunotherapy (Zimberelimab) for 13 cycles and ARM 3: treatment with Sacituzumab Govitecan and Zimberelimab for 8 cycles and Zimberelimab monotherapy for 5 cycles.

The primary objective is to evaluate the disease-free survival (DFS): defined as the length of time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time.

Patient accrual is expected to be completed within 2 years, treatment is planned to extend during 1 years and the patients will be followed up for 2 years. The study will end once survival follow-up has concluded.

DETAILED DESCRIPTION:
This is an open-label, phase III, randomized, stratified (PDL1- vs PDL1+), 3 arms, multicenter clinical trial.

Patients stage IB to IIIA-IIIB (T3N2) after surgical resection if they did not achieve a pathological com-plete response (pCR) will be randomized 1:1:1 to:

* ARM 1: Observational Arm for 10 months
* ARM 2: Immunotherapy (Zimberelimab) treatment for 13 cycles, Q3W
* ARM 3: Sacituzumab Govitecan + Zimberelimab Q3W for 8 cycles + Zimberelimab Q3W for 5 cycles. Patients will receive 8 cycles of the combination and 5 cycles of Zimberelimab monotherapy.

The primary objective is to evaluate the disease-free survival (DFS): defined as the length of time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time.

Disease Free survival (DFS): The time from random assignment to cancer recurrence or death from any cause.

Secondary objectives:

* Overall survival (OS): at 12, 24 and 36 months after the start of adjuvant treatment
* Safety and tolerability of the combination of Sacituzumab Govitecan + Zimberelimab according to CTCAE v5.0.

Exploratory objectives

- To evaluate whether there is a significant association between change in levels of ctDNA between baseline and after adjuvant treatment and OS and DFS.

The total trial duration will be 7 years approximately. Approval-start up: 4-6 months. Patient accrual is expected to be completed within 2 years. One year of treatment and 3 years of follow up, and close-out: 4-6 months. The study will end once survival follow-up has concluded

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients diagnosed of primary non-small cell lung cancer, histologically confirmed.
* 2. Patients should be classified postoperatively in stage IB, IIA, IIB, IIIA or IIIB (N2) according to pathological criteria (pTNM) and according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology
* 3. Complete surgical resection (R0) of the primary NSCLC is also essential. Surgeons are strongly advised to dissect or obtain samples of all accessible lymph node levels, as established in the European Society of Thoracic Surgeons guide. Consequently, at the end of the surgical intervention it is recommended to have obtained samples of a minimum of 3 specific mediastinal ganglionic lobe stations (N2), one of which should include station 7, and at least one N1 station
* 4. The surgical intervention may consist of a lobectomy, sleeve resection, bilobectomy or pneumonectomy, as determined by the responsible surgeon based on intraoperative findings. Patients who have had only segmentectomies or wedge resections are not considered eligible for participation in this study except if R0 resection can be confirmed.
* 5. Only patients that do not achieve pathological complete response (pCR) seen in the surgical piece after neoadjuvant therapy are eligible.
* 6. Preoperative (neoadjuvant) use of platinum-based chemotherapy + immunotherapy (anti PD-1) is mandatory.
* 7. Preoperative, postoperative, or scheduled radiation therapy is not accepted for a later time. Patients with only N2 disease, who have to receive post-operative adjuvant radiotherapy will not be eligible.
* 8. A minimum of 3 weeks must have elapsed between the surgical intervention performed for the NSCLC and the randomization. Adjuvant treatment must start between the 3rd and the 10th week from surgery.
* 9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* 10. Patients aged ≥ 18 years.
* 11. PDL1 value analysed locally (hospital must be able to provide this value before randomization)
* 12. PET-CT and brain CT before randomization to confirm the absence of distant disease.
* 13. Adequate hematologic and organ function
* 14.All patients are notified of the investigational nature of this study and signed a written in-formed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
* 15.For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception
* 16. For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception
* 17. Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs.
* 18.Women who are not postmenopausal or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug.
* 19.Patient capable of proper therapeutic compliance and accessible for correct follow-up
* 20. Patients with a life expectancy of at least more than 12 weeks

Exclusion Criteria:

* 1. Patients with a history of other malignant diseases, with the exception of the following:

  * properly treated non-melanotic skin cancer
  * cancer in situ treated with curative intent or other malignancies treated with curative intent and without signs of disease for a period of> 3 years after the end of the treatment and which, in the opinion of the doctor in charge of their treatment, do not present a substantial risk of relapse of the previous malignant disease.
* 2.T4 patients with invasion of heart, great vessels, carina, trachea, oesophagus or spine
* 3. Patients with ALK translocation, STK11 o KEAP1 known mutations before inclusion in this trial.
* 4. Patients with adenocarcinoma NSCLC must be tested for the common EGFR mutations before inclusion. Patients with any known EGFR mutation cannot be enrolled in the study.
* 5. Patients with a combination of microcytic and non-small cell lung cancer, a carcinoid lung tumor or large cell neuroendocrine carcinoma
* 6. Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of randomization.
* 7. Patients that received live attenuated vaccines within 30 days prior to randomization
* 8. History of a primary immunodeficiency, history of organ allogeneic transplantation, use of immunosuppressive drugs within 28 days before randomization or previous history of toxicity of severe immune mechanism (grade 3 or 4) with other immunological treatments
* 9. Patients with active or uncontrolled infections or with serious medical conditions or disorders that may not allow patient management as established in the protocol.
* 10. Patients who have suffered untreated and / or uncontrolled cardiovascular disorders and / or who have symptomatic cardiac dysfunction
* 11. Pregnant or breastfeeding women
* 12. Patients in whom R0 resection cannot be confirmed.
* 13. Patients with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* 14.Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
* 15. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.
* 16. History of allergy or hypersensitivity to any of the study drug components
* 17. Pleural or pericardial effusion, both will be considered indicative of metastatic disease unless proven otherwise. Patients with pleural effusion not visible on chest-X-ray or too small to perform diagnostic puncture safely may be included.
* 18. Have known history of HIV-1 or 2 with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
* 19.Severe infections within 4 weeks prior to be included in the study, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
* 20.Patients with medical, mental, neurological or psychological condition which in the opinion of the investigator would not permit the patient to understand the patient information sheet or comply with study procedures.
* 21. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder; any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement; or prior pneumonectomy.
* 22. Treatment with systemic immunosuppressive medications
* 23.Patients with uncontrolled comorbidities that may affect the clinical trial compliance.
* 24.Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2031-11-30 (Estimated); Study Completion 2031-11-30 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | The time from random assignment to cancer recurrence or death from any cause, assessed up to 36 months
  Defined as the length of time from randomization to the earliest event defined as disease recurrence, any new lung cancer (even in the opposite lung), or death from any cause at any known point in time.

SECONDARY OUTCOMES:
Overall survival | To evaluate at 12, 24 and 36 months after the start of adjuvant treatment
  defined as the length of time from either the date of diagnosis or the start of the treatment that patients diagnosed with the disease are still alive.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 180 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

OTHER OUTCOMES:
Change in levels of ctDNA during treatment | To analyze at pretreatment, after 6 months of treatment, and at disease relapse, assessed up to 36 months
  Analyze plasma samples and quantifying the amount of circulating tumor DNA (ctDNA) by NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Fundacion GECP
Locations (30):
- Spain (30):
  - Hospital General de Elche, Elche, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Jerez De La Frontera, Jerez de la Frontera, Cádiz
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitari de Gran Canària Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital de Son Espases, Palma de Mallorca, Mallorca
  - Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Clínic De Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital De Basurto, Bilbao
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Santa María Nai, Ourense
  - Hospital Universitari Son Llatzer, Palma de Mallorca
  - Hospital Universitario Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora La Candelaria, Santa Cruz de Tenerife
  - Hospital Virgen del Rocío, Seville
  - Consorci Sanitari de Terrassa, Terrassa
  - Hospital Clínico de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org